CLINICAL TRIAL: NCT02395731
Title: Comprehensive Home-based Dementia Care Coordination for Medicare-Medicaid Dual Eligibles in Maryland
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Jewish Community Services (Other); Johns Hopkins Home Care Group (Unknown); Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00054802
Record Dates: First submitted 2015-03-10; First posted 2015-03-24 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Dementia; Caregiver Burden
Keywords: dual eligible; care coordination; community-based; care quality; care needs; health services; care management; low income; Neuropsychiatric behaviors
MeSH Terms: conditions — Dementia; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MIND at Home- Plus Intervention (Experimental): MIND at Home-Plus is a home-based, care coordination that focuses on persons with dementia living at home and their family caregivers. Its goal is to help persons age in place safely while increasing quality of life. Delivered over 18 months, MIND-Plus systematically assesses and addresses unmet care needs of persons with dementia and their caregivers which are known to be linked to poor health and quality of life outcomes, and that put people at risk for long term care placement. The needs addressed in the MIND program cover a wide range of care domains, ranging from home and medication safety, to cognitive and behavior symptoms management, meaningful activities and legal considerations. The care team made up of a memory care coordinator, nurse, occupational therapist, and physician.
  Interventions: Behavioral: MIND at Home-Plus Intervention

INTERVENTIONS:
Behavioral: MIND at Home-Plus Intervention — MIND at Home-Plus is a home-based, care coordination that focuses on persons with dementia living at home and their family caregivers. Its goal is to help persons age in place safely while increasing quality of life. Delivered over 18 months, MIND-Plus systematically assesses and addresses unmet care needs of persons with dementia and their caregivers which are known to be linked to poor health and quality of life outcomes, and that put people at risk for long term care placement. The needs addressed in the MIND program cover a wide range of care domains, ranging from home and medication safety, to cognitive and behavior symptoms management, meaningful activities and legal considerations. The care team made up of a memory care coordinator, nurse, occupational therapist, and physician.
  Other Names: MIND-Plus

SUMMARY:
This Center for Medicare and Medicaid funded health care innovation award will implement the MIND at Home dementia care coordination program (called MIND at Home-Plus) through two community-based service agencies (Jewish Community Services, Johns Hopkins Home Care Group) to rapidly improve the ability of 600 dually eligible older adults with dementia in the Baltimore region to remain at home while improving care quality, enhancing quality of life, and reducing total health care costs. MIND at Home participants receive an in-home needs assessment followed by up to 18 months of care coordination aimed at filling unmet needs.

DETAILED DESCRIPTION:
The demonstration project has 3 major tasks which will be implemented in concurrent, iterative phases: (1) implement MIND-Plus in 2 community-based health service agencies to rapidly improve the ability of 600 community-living dually eligible older adults with AD in the Baltimore region to remain at home while improving care quality, enhancing quality of life, and reducing total health care costs associated with institutional care or hospitalization; (2) develop a replicable model for nationwide diffusion of the MIND program through a web-based certification package designed to prepare for implementation, build work-force capacity through training certification modules, and provide automated self-monitoring and quality improvement tools; and (3) develop and test a detailed payment model that takes a blended approach and includes provider care management fees with provider performance incentives from division of shared savings.

The investigators hypothesize that the MIND-Plus dementia care coordination program will (1) rapidly improve health & care quality and reduce total health care costs among Medicare-Medicaid dually eligible community-living older adults with AD, (2) drive health care system transformation by creating a new CMS financed benefit that would shift the hub of dementia care coordination to well-trained, dementia competent, interdisciplinary teams based in community health agencies, (3) achieve a sustainable payment model that produces significant net savings and incentives provider performance. This "shovel ready" community-based model is expected to improve outcomes within 6 months and save an estimated net-saving of $12.5 million by over 3 years.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of dementia
* community living
* has identified study partner willing to participate
* english speaking

Exclusion Criteria:

* situation at time of referral is a medical or mental health crisis
* they plan to move out to another area or into a residential care facility in the next 6 months
* they are currently on hospice.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Net cost offset (Medicare and Medicaid costs) of intervention | 18 months
  Estimated per beneficiary per year (PBPY) cost-offset of the MIND at Home-Plus program dementia care coordination program. Defined as the net financial benefit of the program to Medicare and Medicaid expenditures and calculated as the difference in the sum of all Medicare,Medicaid, and intervention costs between intervention group and the sum of all Medicare and Medicaid costs in matched comparison group from (baseline-18 months), adjusted from prior expenditures in the two year period prior to enrollment in the service program or selection into the comparison group.

SECONDARY OUTCOMES:
Change in patient quality of life at 18 months | baseline to 18 months
  Repeated measures within subject data. Person with dementia quality of life as measured by Quality of Life in Alzheimer's Disease (QOL-AD).
Change in caregiver quality of life at 18 months | baseline to 18 months
  Repeated measures within subject data. Caregiver quality of life measured with SF-12
Change in patient unmet dementia-related care needs | baseline to 18 months
  Repeated measures within subject data. Person with dementia unmet care needs as measured by the Johns Hopkins Dementia Care Needs Assessment 2.0
Change in caregiver unmet dementia-related care needs | baseline to 18 months
  Repeated measures within subject data. Family caregiver unmet care needs as measured by the Johns Hopkins Dementia Care Needs Assessment 2.0
Time to long term care placement or death | 18 months
  Time to long term care placement or death for dually eligible persons with dementia compared to a similar matched control group. Kaplan-Meier survival curves will be constructed for each group and adjusted Cox proportional hazards model will be used to assess between-group survival differences.
Time to long term care placement or death | 24 months
  Time to long term care placement or death for dually eligible persons with dementia receiving the MIND intervention compared to a similar matched control group. Kaplan-Meier survival curves will be constructed for each group and adjusted Cox proportional hazards model will be used to assess between-group survival differences.
Change in neuropsychiatric behavior symptoms at 18 months | baseline to 18 months
  Repeated measures within subject data. Neuropsychiatric behavior measured by the Neuropsychiatry Inventory Questionnaire (NPI-Q).
Hospitalization rates | 18 months
  Hospitalization rates for dually eligible persons with dementia receiving the MIND intervention compared to a similar matched control group.
30 day re-hospitalization rates | 18 months
  30 day re-hospitalization rates for dually eligible persons with dementia receiving the MIND intervention compared to a similar matched control group.
Emergency department rates | 18 months
  ED visit rates for dually eligible persons with dementia receiving the MIND intervention compared to a similar matched control group.
Change in patient depression at 18 months | baseline to 18 months
  Repeated measures within subject data. Participant depression measured by Neuropsychiatric Inventory (NPI) section E. Dysphoria.
Change in caregiver depression at 18 months | baseline to 18 months
  Caregiver depression measured by the PHQ-9.
Change in caregiver subjective burden at 18 months | baseline to 18 months
  Repeated measures within subject data. Caregiver burden as measured by objective items (time spent doing activities) and subjective scale (Zarit Burden Interview)
Change in caregiver objective burden at 18 months | baseline to 18 months
  Repeated measures within subject data. Caregiver burden as measured by objective items (time spent doing activities) and subjective scale (Zarit Burden Interview)

OTHER OUTCOMES:
Intervention acceptability | 18 months
  Acceptability as measured by a family caregiver service satisfaction questionnaire at 18 months
Provider satisfaction | 3 years
  MIND care team provider satisfaction as measured by modified STEPPS attitudes toward teamwork questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Quincy Samus, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Samus QM, Davis K, Willink A, Black BS, Reuland M, Leoutsakos J, Roth DL, Wolff J, Gitlin LN, Lyketsos CG, Johnston D. Comprehensive home-based care coordination for vulnerable elders with dementia: Maximizing Independence at Home-Plus-Study protocol. Int J Care Coord. 2017 Dec;20(4):123-134. doi: 10.1177/2053434517744071. Epub 2017 Dec 14. PMID 29607051